CLINICAL TRIAL: NCT01077973
Title: Evaluation Of The Efficacy Of A Novel Ibuprofen Formulation In The Treatment Of Episodic Tension-Type Headache
Brief Title: Study Evaluating A Novel Ibuprofen Formulation In Episodic Tension-Type Headache
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-09-11
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Pain
Keywords: Headache
MeSH Terms: conditions — Pain; Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: Novel Ibuprofen
- Treatment B (Active Comparator)
  Interventions: Drug: Standard Ibuprofen
- Treatment C (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Novel Ibuprofen — Single-dose of novel ibuprofen (equal to 400 mg ibuprofen) plus placebo
  Arms: Treatment A
Drug: Standard Ibuprofen — Single-dose of standard ibuprofen (400mg) plus placebo
  Arms: Treatment B
Drug: Placebo — Single-dose of placebo
  Arms: Treatment C

SUMMARY:
This study will compare the ability of a single-dose of a novel ibuprofen formulation to relieve pain compared to placebo and standard ibuprofen in the treatment of episodic tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years to 65 years of age
* A diagnosis of an episodic tension-type headache, as defined by the International Headache Society
* A history of episodic tension-type headache with the following characteristics: 4 headache episodes per month for the last 6 months of moderately severe intensity; headache generally lasts more than 3 hours if left untreated; adequate headache relief is generally obtained with over-the-counter (OTC) doses of OTC analgesics

Exclusion Criteria:

* Pregnancy or breast-feeding
* Alcohol or substance abuse
* Any serious medical or psychiatric disorder
* History of stomach ulcers, stomach bleed, or other bleeding disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Jayawardena S, Leyva R, Kellstein D. Safety of a novel formulation of ibuprofen sodium compared with standard ibuprofen and placebo. Postgrad Med. 2015 Jan;127(1):33-7. doi: 10.1080/00325481.2015.993268. Epub 2014 Dec 15. PMID 25526232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AH-09-11&StudyName=Study%20Evaluating%20A%20Novel%20Ibuprofen%20Formulation%20In%20Episodic%20Tension-Type%20Headache

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen [Motrin ibuprofen (IB)] 200 milligram (mg) tablet along with single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 mg tablet.
- Ibuprofen Sodium: Single oral dose of 2 ibuprofen sodium 256 mg tablets, equivalent to 400 mg ibuprofen along with single oral dose of 2 placebo tablets matched to ibuprofen (Motrin IB) 200 mg tablet.
- Ibuprofen (Motrin IB): Single oral dose of 2 ibuprofen (Motrin IB) 200 mg tablets (total dose to 400 mg ibuprofen) along with single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 mg tablet.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Started | 41 | 79 | 80
Completed | 41 | 79 | 80
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB) | Total
Number analyzed (Participants) | 41 | 79 | 80 | 200
Age Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (13.5) | 43.4 (13.3) | 40.9 (14.0) | 42.3 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 55 | 55 | 138
  Male | 13 | 24 | 25 | 62
Number of Participants with Pain Severity Score [Number; unit: Participants] — Pain severity score was assessed on a 4-point categorical scale. Total possible pain severity score range was 0 to 3, where 0 = none, 1 = mild, 2 = moderately severe and 3 = severe.
  Participants
    Moderately severe | 30 | 58 | 59 | 147
    Severe | 11 | 21 | 21 | 53

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference From 0-3 Hours (SPRID 0-3) for Ibuprofen Sodium Versus Placebo Tablet
Description: SPRID:time-weighted sum of pain relief rating combined with pain intensity difference (PRID) over 3 hours. SPRID score range:-3 (worst) to 21 (best) for SPRID 0-3. PRID: sum of pain intensity differences (PID) and pain relief rating(PRR) at each time point. PRID score range: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3 (best). PRR:assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 3 hours
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 41 | 79
Units on a scale | 11.2 (4.9) | 10.8 (5.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium-placebo) and 95 percent (%) confidence interval (CI): based on LS means from analysis of variance (ANOVA). Type I error was controlled at 0.05 significance level (2-sided) by stating pair wise comparisons significant only if overall treatment effect among 3 treatment groups was significant and testing in a sequential order Ibuprofen sodium versus (vs.) placebo for SPRID 0-3 then Ibuprofen sodium vs. Ibuprofen (Motrin IB) for time to meaningful relief; Test type: Superiority or Other; p = 0.299, ANOVA — p-value was calculated using ANOVA model with treatment, baseline Pain Severity Rating (PSR), gender and treatment-by-baseline PSR terms; Least-square (LS) mean difference = -1.12, 95% CI 2-sided [-3.23 to 1.00]

2. Primary Outcome: Time to Onset of Meaningful Relief for Ibuprofen Sodium Versus Ibuprofen (Motrin IB) Tablet
Description: Participants evaluated the time to meaningful relief by stopping a second stopwatch labeled 'meaningful relief' at the moment the participant first began to experience meaningful relief. It was also considered achieved if the participant stated "meaningful relief" at the time the first stopwatch was depressed. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 79 | 80
Minutes | 50.3 [41.0 to 60.9] | 55.5 [47.7 to 60.1]
Statistical Analysis 1: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); Hazard Ratio (HR) and corresponding 95% CI were calculated based on the Wald statistic from the proportional hazards (PH) model. Type I error was controlled at 0.05 significance level (2-sided) by stating pair wise comparisons significant only if overall treatment effect among 3 treatment groups was significant and testing in a sequential order Ibuprofen sodium vs. placebo for SPRID 0-3 then Ibuprofen sodium vs. Ibuprofen (Motrin IB) for time to meaningful relief; Test type: Superiority or Other; p = 0.193, Proportional hazards model — p-value was calculated using the PH model with treatment, baseline PSR, gender, and treatment-by-baseline terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.52 to 1.14]

3. Secondary Outcome: Time to Onset of Meaningful Relief: Remaining Comparisons
Description: as for outcome 2
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Minutes | 48.2 [42.7 to 59.8] | 50.3 [41.0 to 60.9] | 55.5 [47.7 to 60.1]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.304, Proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.50 to 1.24]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.936, Proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.65 to 1.59]

4. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief by stopping a stopwatch labeled 'first perceptible relief' at the moment the participant first began to experience any relief. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered. First perceptible relief was considered confirmed by meaningful relief if the participant achieved both "first perceptible" and "meaningful" relief by either depressing the second stopwatch or by indicating that his/her "first perceptible" relief was also "meaningful".
Time Frame: 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Minutes | 42.3 [34.9 to 45.1] | 41.7 [33.5 to 51.3] | 43.8 [36.1 to 51.0]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.072, Proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.41 to 1.04]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.652, Proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.58 to 1.41]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model; Test type: Superiority or Other; p = 0.108, Proportional hazards model — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.49 to 1.07]

5. Secondary Outcome: Pain Relief Rating (PRR)
Description: PRR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  1 hour | 1.9 (1.0) | 1.9 (1.2) | 1.6 (1.0)
  2 hours | 2.6 (1.1) | 2.5 (1.2) | 2.4 (1.2)
  3 hours | 3.0 (1.2) | 2.8 (1.3) | 2.7 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.402, ANOVA — p-value was calculated using ANOVA which was adjusted for treatment, baseline PSR, gender, and treatment-by-baseline terms. Statistical testing was done at 5% significance level (2-sided); LS mean difference = -0.19, 95% CI 2-sided [-0.65 to 0.26]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.407, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.19, 95% CI 2-sided [-0.64 to 0.26]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.991, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.00, 95% CI 2-sided [-0.38 to 0.37]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.313, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.25, 95% CI 2-sided [-0.75 to 0.24]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.621, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.12, 95% CI 2-sided [-0.62 to 0.37]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.533, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.13, 95% CI 2-sided [-0.54 to 0.28]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.352, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.25, 95% CI 2-sided [-0.79 to 0.28]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.573, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.15, 95% CI 2-sided [-0.69 to 0.38]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.657, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.10, 95% CI 2-sided [-0.54 to 0.34]

6. Secondary Outcome: Pain Intensity Difference (PID)
Description: PID was derived by subtracting the pain severity score at a given post-dosing time point [pain severity score range 0 (none) to 3 (severe)] from the baseline score [Baseline pain severity score range 2 (moderately severe) to 3 (severe)]. Total possible score range for PID: -1 (worst) to 3 (best).
Time Frame: 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  1 hour | 0.9 (0.6) | 0.9 (0.6) | 0.8 (0.6)
  2 hours | 1.3 (0.7) | 1.3 (0.7) | 1.2 (0.8)
  3 hours | 1.5 (0.8) | 1.5 (0.9) | 1.4 (0.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.382, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.11, 95% CI 2-sided [-0.36 to 0.14]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.242, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.15, 95% CI 2-sided [-0.39 to 0.10]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.720, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = 0.04, 95% CI 2-sided [-0.17 to 0.24]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.235, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.16, 95% CI 2-sided [-0.43 to 0.11]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.630, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.07, 95% CI 2-sided [-0.34 to 0.20]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.393, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.10, 95% CI 2-sided [-0.32 to 0.13]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.382, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.14, 95% CI 2-sided [-0.46 to 0.18]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; p = 0.995, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = 0.00, 95% CI 2-sided [-0.32 to 0.32]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.287, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.14, 95% CI 2-sided [-0.41 to 0.12]

7. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference (PRID)
Description: PRID was sum of PID and PRR at each post-dosing time point. The overall possible score range, for PRID was -1 (worst) to 7 (best). PID was derived by subtracting the pain severity score at a given post-dosing time point [pain severity score range 0 (none) to 3 (severe)] from the baseline score [Baseline pain severity score range 2 (moderately severe) to 3 (severe)]. Total possible score range for PID: -1 (worst) to 3 (best). PRR was assessed on 5-point categorical pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  1 hour | 2.8 (1.5) | 2.8 (1.8) | 2.4 (1.5)
  2 hours | 3.9 (1.7) | 3.7 (1.9) | 3.6 (1.9)
  3 hours | 4.5 (2.0) | 4.3 (2.1) | 4.1 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.377, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.30, 95% CI 2-sided [-0.98 to 0.37]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p = 0.324, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.34, 95% CI 2-sided [-1.01 to 0.34]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.902, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = 0.03, 95% CI 2-sided [-0.52 to 0.59]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 4]; Test type: Superiority or Other; p = 0.273, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.42, 95% CI 2-sided [-1.17 to 0.33]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.616, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.19, 95% CI 2-sided [-0.94 to 0.56]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 6]; Test type: Superiority or Other; p = 0.471, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-0.85 to 0.39]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.356, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.40, 95% CI 2-sided [-1.24 to 0.45]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 8]; Test type: Superiority or Other; p = 0.722, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.15, 95% CI 2-sided [-1.00 to 0.69]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 5, analysis 9]; Test type: Superiority or Other; p = 0.493, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.24, 95% CI 2-sided [-0.94 to 0.46]

8. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID)
Description: SPID: time-weighted sum of PID over 2 and 3 hours. SPID score range was -2(worst) to 6 (best) for SPID 0-2 and -3 (worst) to 9 (best) for SPID 0-3. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3 (best).
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  SPID 0-2 | 2.2 (1.3) | 2.2 (1.3) | 2.0 (1.3)
  SPID 0-3 | 3.8 (2.0) | 3.6 (2.1) | 3.4 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.259, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.27, 95% CI 2-sided [-0.75 to 0.20]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); SPID 0-2: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.378, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.21, 95% CI 2-sided [-0.69 to 0.26]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPID 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.762, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.06, 95% CI 2-sided [-0.45 to 0.33]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; SPID 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.281, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.42, 95% CI 2-sided [-1.17 to 0.34]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); SPID 0-3: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.582, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.21, 95% CI 2-sided [-0.97 to 0.55]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPID 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.523, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.20, 95% CI 2-sided [-0.83 to 0.42]

9. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR)
Description: TOTPAR: time-weighted sum of PRR over 2 and 3 hours. TOTPAR score range was 0 (worst) to 8 (best) for TOTPAR 0-2 and 0 (worst) to 12 (best) for TOTPAR 0-3. PRR was assessed on a 5-point categorical pain relief rating scale wherein 0=No relief to 4=Complete relief.
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  TOTPAR 0-2 | 4.5 (2.0) | 4.4 (2.3) | 4.1 (2.0)
  TOTPAR 0-3 | 7.5 (3.1) | 7.2 (3.5) | 6.8 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.327, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.45, 95% CI 2-sided [-1.35 to 0.45]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); TOTPAR 0-2: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.489, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.32, 95% CI 2-sided [-1.21 to 0.58]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); TOTPAR 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.726, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.13, 95% CI 2-sided [-0.88 to 0.61]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; TOTPAR 0-3: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.320, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.70, 95% CI 2-sided [-2.09 to 0.69]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); TOTPAR 0-3: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.506, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.47, 95% CI 2-sided [-1.86 to 0.92]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); TOTPAR 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.691, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.23, 95% CI 2-sided [-1.38 to 0.92]

10. Secondary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference (SPRID)
Description: SPRID: time-weighted sum of PRID over 2 and 3 hours. SPRID score range was -2(worst) to 14(best) for SPRID 0-2 and -3 (worst) to 21 (best) for SPRID 0-3. PRID: sum of PID and PRR at each time point. Total score range for PRID: -1=worst to 7=best. PID: baseline pain severity score minus pain severity score at a given time point (score range 0=none to 3=severe; baseline score range 2=moderately severe to 3=severe). Total score range for PID: -1(worst) to 3(best), PRR: assessed on 5-point pain relief rating scale (0=No relief to 4=Complete relief).
Time Frame: 0 to 2, 0 to 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Units on a scale
  SPRID 0-2 | 6.7 (3.1) | 6.5 (3.4) | 6.1 (3.2)
  SPRID 0-3 | 11.2 (4.9) | 10.8 (5.3) | 10.2 (5.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; SPRID 0-2: Treatment difference (Ibuprofen sodium - placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.292, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.72, 95% CI 2-sided [-2.07 to 0.62]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); SPRID 0-2: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.439, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.53, 95% CI 2-sided [-1.87 to 0.82]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPRID 0-2: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.733, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.19, 95% CI 2-sided [-1.31 to 0.92]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen (Motrin IB); SPRID 0-3: Treatment difference [Ibuprofen (Motrin IB) - placebo] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.526, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.68, 95% CI 2-sided [-2.80 to 1.43]
Statistical Analysis 5: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); SPRID 0-3: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.624, ANOVA — [p-value comment as in outcome 5, analysis 1]; LS mean difference = -0.44, 95% CI 2-sided [-2.19 to 1.31]

11. Secondary Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief evaluated by stopping a second stopwatch labeled 'meaningful relief' at the moment the participant first began to experience meaningful relief. It was also considered achieved if the participant stated "meaningful relief" at the time the first stopwatch was depressed. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered.
Time Frame: 0.5, 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Percentage of participants
  0.5 hours | 14.6 | 17.7 | 10.0
  1 hour | 65.9 | 58.2 | 60.0
  2 hours | 85.4 | 79.7 | 81.3
  3 hours | 85.4 | 81.0 | 82.5
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.672, Cochran-Mantel-Haenszel — p-value was calculated using CMH test which was adjusted for baseline PSR, and gender. Statistical testing was done at 5% significance level (2-sided); Difference in proportion = 3.02, 95% CI 2-sided [-11.03 to 17.07]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); 0.5 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.467, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -4.47, 95% CI 2-sided [-17.61 to 8.68]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 0.5 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.164, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 7.55, 95% CI 2-sided [-2.96 to 18.05]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.427, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -7.52, 95% CI 2-sided [-25.96 to 10.92]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.537, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -5.66, 95% CI 2-sided [-23.57 to 12.25]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 1 hour: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.813, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -1.83, 95% CI 2-sided [-16.88 to 13.22]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.455, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -5.50, 95% CI 2-sided [-19.24 to 8.24]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.570, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -4.02, 95% CI 2-sided [-17.63 to 9.59]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 2 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.792, Cochran-Mantel-Haenszel — p-value was calculated using CMH test which was adjusted which was adjusted for baseline PSR, and gender. Statistical testing was done at 5% significance level (2-sided); Difference in proportion = -1.65, 95% CI 2-sided [-13.80 to 10.50]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; 3 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.556, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -4.25, 95% CI 2-sided [-17.82 to 9.33]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen (Motrin IB) - placebo] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.689, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -2.77, 95% CI 2-sided [-16.24 to 10.69]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); 3 hours: Treatment difference [Ibuprofen sodium - Ibuprofen (Motrin IB)] and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.786, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -1.65, 95% CI 2-sided [-13.45 to 10.14]

12. Secondary Outcome: Cumulative Percentage of Participants With Confirmed First Perceptible Relief
Description: Percentage of participants with first perceptible relief evaluated by stopping a stopwatch labeled 'first perceptible relief' at the moment the participant first began to experience any relief. Stopwatch was active up to 3 hours after dosing or until stopped by the participant, or rescue medication was administered. First perceptible relief was considered confirmed by meaningful relief if the participant achieved both "first perceptible" and "meaningful" relief by either depressing the second stopwatch or by indicating that his/her "first perceptible" relief was also "meaningful".
Time Frame: 0.5, 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Percentage of participants
  0.5 hours | 24.4 | 30.4 | 28.8
  1 hour | 80.5 | 67.1 | 72.5
  2 hours | 85.4 | 81.0 | 82.5
  3 hours | 85.4 | 81.0 | 82.5
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.480, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 6.06, 95% CI 2-sided [-10.86 to 22.99]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 2]; Test type: Superiority or Other; p = 0.612, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 4.34, 95% CI 2-sided [-12.55 to 21.23]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.839, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 1.47, 95% CI 2-sided [-12.60 to 15.55]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.130, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -13.20, 95% CI 2-sided [-29.40 to 2.99]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p = 0.331, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -7.83, 95% CI 2-sided [-23.39 to 7.73]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.450, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -5.50, 95% CI 2-sided [-19.59 to 8.59]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.556, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -4.25, 95% CI 2-sided [-17.82 to 9.33]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 8]; Test type: Superiority or Other; p = 0.689, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -2.77, 95% CI 2-sided [-16.24 to 10.69]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; p = 0.786, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -1.65, 95% CI 2-sided [-13.45 to 10.14]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p = 0.556, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -4.25, 95% CI 2-sided [-17.82 to 9.33]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.689, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -2.77, 95% CI 2-sided [-16.24 to 10.69]
Statistical Analysis 12: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 12]; Test type: Superiority or Other; p = 0.786, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -1.65, 95% CI 2-sided [-13.45 to 10.14]

13. Secondary Outcome: Time to Treatment Failure
Description: Median time of dropping out of the participants from the study due to lack of efficacy or received rescue medication, whichever came first.
Time Frame: 0 to 3 hours
Population: Data was not analyzed as there were no treatment failures observed and no participant received rescue medication in the study.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Percentage of participants who withdrew from the study due to lack of efficacy or received rescue medication.
Time Frame: 0 to 3 hours
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Cumulative Percentage of Participants With Complete Relief
Description: Complete relief was defined as a PRR of 4. PRR was assessed on a 5-point categorical pain relief rating scale where 0=No relief to 4=Complete relief.
Time Frame: 1, 2, 3 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Number analyzed (Participants) | 41 | 79 | 80
Percentage of participants
  1 hour | 2.4 | 6.3 | 1.3
  2 hours | 17.1 | 21.5 | 15.0
  3 hours | 41.5 | 40.5 | 35.0
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 4]; Test type: Superiority or Other; p = 0.355, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 3.89, 95% CI 2-sided [-3.33 to 11.10]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 5]; Test type: Superiority or Other; p = 0.623, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -1.21, 95% CI 2-sided [-6.62 to 4.20]
Statistical Analysis 3: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 6]; Test type: Superiority or Other; p = 0.094, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 5.10, 95% CI 2-sided [-0.90 to 11.11]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 7]; Test type: Superiority or Other; p = 0.565, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 4.43, 95% CI 2-sided [-10.43 to 19.29]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 8]; Test type: Superiority or Other; p = 0.765, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -2.09, 95% CI 2-sided [-16.15 to 11.97]
Statistical Analysis 6: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 9]; Test type: Superiority or Other; p = 0.288, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 6.47, 95% CI 2-sided [-5.43 to 18.37]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 11, analysis 10]; Test type: Superiority or Other; p = 0.928, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -0.87, 95% CI 2-sided [-20.00 to 18.27]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 11]; Test type: Superiority or Other; p = 0.495, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = -6.40, 95% CI 2-sided [-25.14 to 12.33]
Statistical Analysis 9: Comparison: Ibuprofen Sodium vs Ibuprofen (Motrin IB); [analysis description as in outcome 11, analysis 12]; Test type: Superiority or Other; p = 0.477, Cochran-Mantel-Haenszel — [p-value comment as in outcome 11, analysis 1]; Difference in proportion = 5.46, 95% CI 2-sided [-9.66 to 20.59]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen Sodium | Ibuprofen (Motrin IB)
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/79 | 0/80
Other Adverse Events (participants affected / at risk) | 0/41 | 0/79 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.